CLINICAL TRIAL: NCT02800603
Title: "Making the Race Fair for Young Children at Risk": A Targeted Prevention Approach to Reducing Child Emotional and Behaviour Problems
Brief Title: A Targeted Prevention Approach to Reducing Child Emotional and Behaviour Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Arizona State University (Other); University of Calgary (Other); Simon Fraser University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FCU
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Emotional Problems; Behavior Problems
Keywords: preschool mental health; emotional and behaviour problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Check Up (Experimental): FCU Intervention: All 280 participants will undergo screening and a baseline FCU assessment before randomization. Once randomized, the FCU group (n=140) will be provided with a feedback visit and up to 6 optional sessions of the EDP curriculum over 16 weeks.
  Interventions: Behavioral: Family Check Up
- Community Control (No Intervention): The Community Control group (n=140) will receive general information that includes a list of all the relevant services available in Hamilton. As such, the community control group would be provided with all the information needed to obtain standard care.

INTERVENTIONS:
Behavioral: Family Check Up — The FCU is an ecologically sensitive, evidence-based, targeted intervention that aims to reduce child EBP. Features of the FCU: 1) Assessment-driven: a multi-method, multi-informant assessment in which the consultant reviews strengths and difficulties across domains of contextual risk, family functioning and child health. A tailored intervention plan is then created based on results 2) Motivational interviewing: Caregivers engage in self-assessment about motivation and barriers to addressing factors that may perpetuate risk. The consultant and caregiver work to establish a menu of services 3) The family may be offered up to 6 sessions of the "Everyday Parenting" curriculum. The FCU has demonstrated effectiveness and cultural sensitivity across multiple US settings.
  Arms: Family Check Up

SUMMARY:
The purpose of the study is to evaluate the first Canadian implementation project of the Family Check up (FCU), an evidence-based prevention and early intervention model that engages families and communities in reducing the burden of childhood emotional and behaviour problems (EBP).

DETAILED DESCRIPTION:
The aim of this study is to establish and evaluate the first Canadian implementation project of the FCU as an evidence-based prevention and early intervention model that engages families and communities in reducing the burden of childhood EBP. These objectives will be achieved in two foundational phases. During Phase 1, the clinical and systems infrastructure required to deliver, sustain and ultimately scale up the FCU will be built. During Phase 2, a 1:1 randomized controlled trial (RCT) will be conducted. The RCT will involve 280 participating caregiver-child dyads to examine the effects of the FCU as a targeted prevention intervention within the Canadian context, as delivered to caregivers and children aged 2-4 years at high risk of persistent childhood EBP.

Phase 1: Training, and Implementation: The REACH Institute at Arizona State University has developed an efficient model for international implementation of the FCU. They will help implement the intervention within McMaster Children's Hospital (MCH), train MCH therapists as FCU consultants, and two trainers. All therapists will be credentialed as FCU consultants by REACH through a process of supervision, consultation and monitoring of therapeutic fidelity.

Phase 2: Investigators will conduct a 1:1 randomized controlled trial of 280 children aged 2-4 years into either the FCU (n=140) or community control (CC, n=140). All 280 participants will undergo screening and a baseline FCU assessment before randomization. Once randomized, the FCU group will be provided with a feedback visit and up to 6 optional sessions of the Everyday Parenting (EDP) curriculum over 16 weeks. The CC group will receive general information about currently available community services in Hamilton. At 6 months, both groups will undergo light assessments. At 12 months both groups will repeat the baseline assessment, and the FCU group will have 1-2 FCU visits.

ELIGIBILITY:
Inclusion Criteria: Screening eligibility criteria include:

1. Custodial caregivers of a child aged 2 years, 0 months to 4 years, 11 months.
2. Definition of "at-risk" for child EBP as measured by (a) OR (b):

   * Elevated child EBP as indexed by above-population mean total scores on Strengths and Difficulties Questionnaire (SDQ), plus one of the following family or contextual risk factors

     * Caregiver challenges: teen parent status, caregiver mental health problems (as indexed by K6 psychological distress scale), lone caregiver
     * Sociodemographic risk factors (as indexed by the 2014 Ontario Child Health Study (OCHS) demographics questionnaire): family income below low-income cut-off (LICO), caregiver with less than grade 12 education, caregiver on social assistance.
   * Families who score within norms on caregiver or sociodemographic risk AND child SDQ scores fall within the "high" range, indicating significant burden of EBP (and thus increased risk of persistent, severe problems over time).
3. Caregivers with sufficient knowledge of English needed for assessment measures
4. Caregivers capable of giving informed, written consent

Exclusion Criteria:

1. Children with suspected severe to profound developmental delay
2. Current enrolment in another clinical intervention trial
3. Caregiver or child with a serious medical condition that, based on Investigator judgment, might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome- Change in Child Externalizing Behaviors | Primary outcome will be measured at baseline, 6- and 12-months after enrollment
  Change in Child Behavior Checklist (CBCL) scores

SECONDARY OUTCOMES:
Secondary Outcome - Change in Parental Mental Health | This will be measured at baseline, 6- and 12-months
  The Kessler-6 (K6) will be used to measure change in psychological distress over time
Secondary Outcome - Change in Parental Stress | This will be measured at baseline and 12-months
  Parenting Daily Hassles will be used to measure changes in parental stress over time
Secondary Outcome - Change in Positive Parenting Practice | This will be measured at baseline and 12-months
  Positive parenting practice will be coded from videotaped parent-child interactions - outcome is change in positive parenting practice over time
Secondary Outcome - Change in Child Compliance | This will be measured at baseline and 12-months
  The Coder Impressions Inventory (COIMP) will be used to score the child's behaviour from videotaped interactions - outcome is change in behaviour over time

OTHER OUTCOMES:
Exploratory outcome - Health Service Utilization | This will be measured at baseline, 3-, 6-, 9- and 12- months.
  Service utilization questionnaire
Exploratory outcome - Change in Behavioural Observations of Parenting | This will be measured at baseline, 6-months and 12 months.
  Behavioural Observations of Parenting will be assessed using videotapes of structured interaction between the child and parent
Exploratory outcome - Change in Parental Emotional Regulation | Exploratory outcomes will be measured at baseline and at 12 months.
  Difficulties in Emotion Regulation Scale (DERS)
Exploratory outcome - Change in Child Emotional Regulation | This will be measured at baseline and at 12 months.
  Child emotional regulation will be assessed using videotapes of the child performing structured tasks
Exploratory outcome -Parent Executive Functioning | This will be measured at baseline.
  Parent executive functioning will be assessed using observation of structured tasks
Exploratory outcome - Change in Child Executive Functioning | This will be measured at baseline and at 12 months.
  Child executive functioning will be assessed using observation of structured tasks
Exploratory outcome - Change in Hair Cortisol | This will be measured at baseline, 6-months and 12 months.
  Small amounts of hair will be collected from child and parents to assess hair cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Bennett, MD/PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egger HL, Angold A. Common emotional and behavioral disorders in preschool children: presentation, nosology, and epidemiology. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):313-37. doi: 10.1111/j.1469-7610.2006.01618.x. PMID 16492262
- [Background] Cadman D, Boyle M, Szatmari P, Offord DR. Chronic illness, disability, and mental and social well-being: findings of the Ontario Child Health Study. Pediatrics. 1987 May;79(5):805-13. PMID 2952939
- [Background] Furniss T, Beyer T, Guggenmos J. Prevalence of behavioural and emotional problems among six-years-old preschool children: baseline results of a prospective longitudinal study. Soc Psychiatry Psychiatr Epidemiol. 2006 May;41(5):394-9. doi: 10.1007/s00127-006-0045-3. Epub 2006 Mar 25. PMID 16565920
- [Background] Skovgaard AM. Mental health problems and psychopathology in infancy and early childhood. An epidemiological study. Dan Med Bull. 2010 Oct;57(10):B4193. PMID 21040689
- [Background] Shonkoff JP, Richter L, van der Gaag J, Bhutta ZA. An integrated scientific framework for child survival and early childhood development. Pediatrics. 2012 Feb;129(2):e460-72. doi: 10.1542/peds.2011-0366. Epub 2012 Jan 4. PMID 22218840
- [Background] Bernier A, Carlson SM, Whipple N. From external regulation to self-regulation: early parenting precursors of young children's executive functioning. Child Dev. 2010 Jan-Feb;81(1):326-39. doi: 10.1111/j.1467-8624.2009.01397.x. PMID 20331670
- [Background] Gill AM, Hyde LW, Shaw DS, Dishion TJ, Wilson MN. The Family Check-Up in early childhood: a case study of intervention process and change. J Clin Child Adolesc Psychol. 2008 Oct;37(4):893-904. doi: 10.1080/15374410802359858. PMID 18991138
- [Background] Smith JD, Knoble NB, Zerr AA, Dishion TJ, Stormshak EA. Family check-up effects across diverse ethnic groups: reducing early-adolescence antisocial behavior by reducing family conflict. J Clin Child Adolesc Psychol. 2014;43(3):400-14. doi: 10.1080/15374416.2014.888670. Epub 2014 Apr 14. PMID 24731120
- [Background] Shaw DS, Dishion TJ, Supplee L, Gardner F, Arnds K. Randomized trial of a family-centered approach to the prevention of early conduct problems: 2-year effects of the family check-up in early childhood. J Consult Clin Psychol. 2006 Feb;74(1):1-9. doi: 10.1037/0022-006X.74.1.1. PMID 16551138
- [Background] Dishion TJ, Shaw D, Connell A, Gardner F, Weaver C, Wilson M. The family check-up with high-risk indigent families: preventing problem behavior by increasing parents' positive behavior support in early childhood. Child Dev. 2008 Sep-Oct;79(5):1395-414. doi: 10.1111/j.1467-8624.2008.01195.x. PMID 18826532
- [Background] Dishion TJ, Brennan LM, Shaw DS, McEachern AD, Wilson MN, Jo B. Prevention of problem behavior through annual family check-ups in early childhood: intervention effects from home to early elementary school. J Abnorm Child Psychol. 2014;42(3):343-54. doi: 10.1007/s10802-013-9768-2. PMID 24022677
- [Background] Connell A, Bullock BM, Dishion TJ, Shaw D, Wilson M, Gardner F. Family intervention effects on co-occurring early childhood behavioral and emotional problems: a latent transition analysis approach. J Abnorm Child Psychol. 2008 Nov;36(8):1211-25. doi: 10.1007/s10802-008-9244-6. PMID 18473160
- [Background] Lunkenheimer ES, Dishion TJ, Shaw DS, Connell AM, Gardner F, Wilson MN, Skuban EM. Collateral benefits of the Family Check-Up on early childhood school readiness: indirect effects of parents' positive behavior support. Dev Psychol. 2008 Nov;44(6):1737-52. doi: 10.1037/a0013858. PMID 18999335
- [Background] Weaver CM, Shaw DS, Crossan JL, Dishion TJ, Wilson MN. Parent-child conflict and early childhood adjustment in two-parent low-income families: parallel developmental processes. Child Psychiatry Hum Dev. 2015 Feb;46(1):94-107. doi: 10.1007/s10578-014-0455-5. PMID 24610382
- [Background] Brennan LM, Shelleby EC, Shaw DS, Gardner F, Dishion TJ, Wilson M. Indirect Effects of the Family Check-Up on School-Age Academic Achievement Through Improvements in Parenting in Early Childhood. J Educ Psychol. 2013 Aug 1;105(3):10.1037/a0032096. doi: 10.1037/a0032096. PMID 24319295
- [Background] Leijten P, Shaw DS, Gardner F, Wilson MN, Matthys W, Dishion TJ. The family check-up and service use in high-risk families of young children: a prevention strategy with a bridge to community-based treatment. Prev Sci. 2015 Apr;16(3):397-406. doi: 10.1007/s11121-014-0479-x. PMID 24643281
- [Background] Shaw DS, Connell A, Dishion TJ, Wilson MN, Gardner F. Improvements in maternal depression as a mediator of intervention effects on early childhood problem behavior. Dev Psychopathol. 2009 Spring;21(2):417-39. doi: 10.1017/S0954579409000236. PMID 19338691
- [Background] Chang H, Shaw DS, Dishion TJ, Gardner F, Wilson MN. Direct and indirect effects of the family check-up on self-regulation from toddlerhood to early school-age. J Abnorm Child Psychol. 2014 Oct;42(7):1117-28. doi: 10.1007/s10802-014-9859-8. PMID 24599383
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Achenbach TM, Ruffle TM. The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatr Rev. 2000 Aug;21(8):265-71. doi: 10.1542/pir.21-8-265. No abstract available. PMID 10922023
- [Background] Willoughby MT, Blair CB, Wirth RJ, Greenberg M. The measurement of executive function at age 5: psychometric properties and relationship to academic achievement. Psychol Assess. 2012 Mar;24(1):226-39. doi: 10.1037/a0025361. Epub 2011 Oct 3. PMID 21966934
- [Background] Mischel W, Shoda Y, Rodriguez MI. Delay of gratification in children. Science. 1989 May 26;244(4907):933-8. doi: 10.1126/science.2658056.
- [Background] Landry SH, Miller-Loncar CL, Smith KE, Swank PR. The role of early parenting in children's development of executive processes. Dev Neuropsychol. 2002;21(1):15-41. doi: 10.1207/S15326942DN2101_2. PMID 12058834
- [Background] Kochanska G, Murray K, Jacques TY, Koenig AL, Vandegeest KA. Inhibitory control in young children and its role in emerging internalization. Child Dev. 1996 Apr;67(2):490-507. PMID 8625724
- [Background] Zelazo PD, Muller U, Frye D, Marcovitch S, Argitis G, Boseovski J, Chiang JK, Hongwanishkul D, Schuster BV, Sutherland A. The development of executive function in early childhood. Monogr Soc Res Child Dev. 2003;68(3):vii-137. doi: 10.1111/j.0037-976x.2003.00260.x. PMID 14723273
- [Background] Gerstadt CL, Hong YJ, Diamond A. The relationship between cognition and action: performance of children 3 1/2-7 years old on a Stroop-like day-night test. Cognition. 1994 Nov;53(2):129-53. doi: 10.1016/0010-0277(94)90068-x. PMID 7805351
- [Background] Carlson SM. Developmentally sensitive measures of executive function in preschool children. Dev Neuropsychol. 2005;28(2):595-616. doi: 10.1207/s15326942dn2802_3. PMID 16144429
- [Background] Russell E, Koren G, Rieder M, Van Uum S. Hair cortisol as a biological marker of chronic stress: current status, future directions and unanswered questions. Psychoneuroendocrinology. 2012 May;37(5):589-601. doi: 10.1016/j.psyneuen.2011.09.009. Epub 2011 Oct 4. PMID 21974976
- [Background] Stalder T, Kirschbaum C. Analysis of cortisol in hair--state of the art and future directions. Brain Behav Immun. 2012 Oct;26(7):1019-29. doi: 10.1016/j.bbi.2012.02.002. Epub 2012 Feb 15. PMID 22366690
- [Background] Manenschijn L, Koper JW, Lamberts SW, van Rossum EF. Evaluation of a method to measure long term cortisol levels. Steroids. 2011 Sep-Oct;76(10-11):1032-6. doi: 10.1016/j.steroids.2011.04.005. Epub 2011 Apr 14. PMID 21515299
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Dumas JE, Nissley J, Nordstrom A, Smith EP, Prinz RJ, Levine DW. Home chaos: sociodemographic, parenting, interactional, and child correlates. J Clin Child Adolesc Psychol. 2005 Mar;34(1):93-104. doi: 10.1207/s15374424jccp3401_9. PMID 15677284
- [Background] Smith JD, Dishion TJ, Shaw DS, Wilson MN. Indirect effects of fidelity to the family check-up on changes in parenting and early childhood problem behaviors. J Consult Clin Psychol. 2013 Dec;81(6):962-74. doi: 10.1037/a0033950. Epub 2013 Jul 29. PMID 23895087
- [Background] Chiapa A, Smith JD, Kim H, Dishion TJ, Shaw DS, Wilson MN. The trajectory of fidelity in a multiyear trial of the family check-up predicts change in child problem behavior. J Consult Clin Psychol. 2015 Oct;83(5):1006-11. doi: 10.1037/ccp0000034. Epub 2015 Jun 29. PMID 26121303
- [Background] Boyle MH, Offord DR, Hofmann HG, Catlin GP, Byles JA, Cadman DT, Crawford JW, Links PS, Rae-Grant NI, Szatmari P. Ontario Child Health Study. I. Methodology. Arch Gen Psychiatry. 1987 Sep;44(9):826-31. doi: 10.1001/archpsyc.1987.01800210078012. PMID 3632257
- [Background] Radloff, L. S. The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement 1(3): 385-401, 1977.
- [Background] Eaton WW, Muntaner C, Smith C, Tien A, Ybarra M. The Use of Psychological Testing for Treatment Planning and Outcomes Assessment, Volume 3: Instruments for Adults, 3rd ed. Mahwah, NJ: Lawrence Erlbaum; 2004. Chapter 11, Center for Epidemiologic Studies Depression Scale: Review and revision (CESD and CESD-R); p 363-377.
- [Background] Gratz, K.L., & Roemer, L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment 26(1): 41-54, 2004.
- [Derived] Bennett T, Georgiades K, Gonzalez A, Janus M, Lipman E, Pires P, Prime H, Duku E, Jambon M, McLennan JD, Gross J; Making the Race Fair Study Team. Targeted Child Mental Health Prevention and Parenting Support Within a Canadian Context: A Randomized Controlled Trial Evaluating the U.S.-Developed Family Check-Up(R). Prev Sci. 2025 May;26(4):555-567. doi: 10.1007/s11121-024-01741-3. Epub 2024 Nov 22. PMID 39572487